CLINICAL TRIAL: NCT05995756
Title: Evaluate the Safety and Efficacy of Sinocare CGM System Regarding Real Time Glucose
Brief Title: Evaluate the Safety and Efficacy of Sinocare CGM System Regarding Real Time Glucose Level Monitoring
Status: Completed | Type: Observational
Sponsor: Sinocare (Industry)
Responsible Party: Sponsor
Other Study IDs: NPI031-CIP-001
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Type 1 or Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In pateint
- Out pateint

SUMMARY:
From Jan 2022 to June 2022, 120 subjects (22-75 years of age, mean ±standard deviation [SD] of 53.20 ±14.49 years) with type 1 or type 2 diabetes participated in the study in P.R. China. Subjects wore two sensors in the abdomen which were paired with smart devices running a glucose monitoring mobile application (i3/H3 CGM APP). Subjects were asked to undergo one in-clinic visit (on one of the study days 2, 7-9, or 15) for 7-hour long YSI frequent sampling test (FST) periods, where intravenous (IV) blood samples were drawn every 15 min and analyzed using the YSI 2300 STAT Plus Glucose & Lactate Analyzer (Yellow Springs Instrument, YSI Life Sciences, Yellow Springs, OH).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years, male or female;
2. Clinically diagnosed with diabetes;
3. Being willing to wear the investigational device for the duration set according to its service life, and conduct glucose monitoring;
4. Consent to participate in this clinical study, and sign the Informed Consent Form (ICF).

Exclusion Criteria:

1. Disagree to wear the investigational device continuously according to the requirements of the trial;
2. Refuse venous blood collection for 7 consecutive hours (every 15 minutes) on a certain day during the trial;
3. Plan to undergo magnetic resonance imaging (MRI) during the clinical trial;
4. With diffuse subcutaneous nodules at the wearing site of the investigational device;
5. Have a history of diabetic ketoacidosis or hyperosmolar hyperglycemic state within the 6 months prior to screening;
6. With mental disorders, lack of self-control and inability to express clearly;
7. Have participated in any other clinical trial within the past 1 month;
8. Where the investigator thinks not suitable for being enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (Aged ≥18) TD1 and TD2
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
overall mean absolute relative difference (MARD) | 8 or 15 days

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Pinggu Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha

IPD SHARING:
Plan to Share IPD: No